CLINICAL TRIAL: NCT03405805
Title: The Establishment of Serotype-specific Immunological Memory Against Pneumococcus by a 3+1 Versus a 2+1 or 3+0 Infant PCV13 Vaccination Schedule
Brief Title: Immunological Memory Against Pneumococcus Induced by 3 Infant PCV 13 Vaccination Schedules
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aghia Sophia Children's Hospital of Athens (Other)
Responsible Party: Principal Investigator, Vana Spoulou, Assistant Professor of Paediatrics, Aghia Sophia Children's Hospital of Athens
Other Study IDs: isppd2018
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Immunogenicity, Vaccine; Immunologic Memory
MeSH Terms: interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 3+1: Healthy infants will receive 4 doses of the 13-valent pneumococcal conjugate vaccine (PCV13) at 2,4,6 and 12 months of age and blood and serum collection pre- dose, 7 days post- (only blood) and 28 days post- last dose.
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine (PCV13)
- 3+0: Healthy infants will receive 3 doses of the 13-valent pneumococcal conjugate vaccine (PCV13) at 2,4 and 6 months of age and blood and serum collection pre- dose, 7 days post- (only blood) and 28 days post- last dose.
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine (PCV13)
- 2+1: Healthy infants will receive 3 doses of the 13-valent pneumococcal conjugate vaccine (PCV13) at 2,4 and 12 months of age and blood and serum collection pre- dose, 7 days post- (only blood) and 28 days post- last dose.
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine (PCV13)

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine (PCV13) — Vaccination with PCV13
  Other Names: Prevenar13

SUMMARY:
The purpose of this study is to evaluate the establishment of immunological memory between the 3 different infant vaccination schedules with the 13-valent pneumococcal conjugate vaccine (PCV13) currently in use. We aim to determine the optimal schedule for the establishment of antigen-specific memory B-cell pool, which may serve as a correlate for longevity of immunological memory against vaccine serotypes. Moreover, we will study the transcriptome profiles expressed by peripheral lymphocytes during each immune response in an attempt to reveal immunological mechanisms beyond the antibody and circulating B cells level.

ELIGIBILITY:
Inclusion Criteria:

* 2-15 months of age

Exclusion Criteria:

* previously recorded allergy to PCV
* intravenous immunoglobulin (IVIG) given within the previous 6 months
* primary or secondary immunodeficiency
* any chronic medical condition

Ages: 2 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy infants 2-15 months of age living in Athens, Greece
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-12-12 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
immunoglobulin G (IgG) antibody serum titers (measured by ELISA) | 28 days post last vaccine dose
  measurement of IgG antibody titers in serum pre- and post- last dose of PCV13
switched immunoglobulin G (swIgG) B memory cell response (measured by flow cytometry) | 28 days post last vaccine dose
  phenotype characterisation of swIgG memory B cells pre- and post- last dose of PCV13
immunoglobulin M (IgM) B memory cell response (measured by flow cytometry) | 28 days post last vaccine dose
  phenotype characterisation of IgM memory B cells pre- and post- last dose of PCV13

SECONDARY OUTCOMES:
Transcriptional profile of Peripheral Blood Mononuclear Cells (PBMC) in response to PCV13 (measured by RNA-Sequencing) | 7 days post last vaccine dose
  transcriptome analysis of PBMCs pre- and post last dose of PCV13 on a cohort of patients

CONTACTS AND LOCATIONS:
Overall Officials: Vana Spoulou, MD, PhD, Study Chair — "Aghia Sophia" Children's Hospital
Locations (1):
- 'Aghia Sophia' Children's Hospital, Athens, Attica, Greece